CLINICAL TRIAL: NCT00576797
Title: Genomic Tools for Studying the Ecology of the Human Vaginal Microflora
Acronym: VM
Status: Completed | Type: Observational
Sponsor: Emory University (Other)
Collaborators: University of Maryland (Other); National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Kevin Ault, MD, Principal Investigator, Emory University
Other Study IDs: IRB00001794; U01AI070921-01 (NIH)
Record Dates: First submitted 2007-12-17; First posted 2007-12-19 (Estimated); Last update posted 2016-02-02 (Estimated); Status verified 2016-02

CONDITIONS: Healthy
Keywords: vaginal; bacteria; microflora; bacterial DNA; To determine the normal bacteria in the vagina

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — vaginal secretions
Oversight: Data Monitoring Committee: No

SUMMARY:
The human vagina contains a large number of normal bacteria. These bacteria are important because provide protection against other bacteria that may cause disease. Several important diseases are linked to abnormal bacteria in the vagina. Women with abnormal bacteria in the vagina are more likely to be infected with human immunodeficiency virus, the virus that causes AIDS. Also women with unusual bacteria in their vagina are more likely to deliver a premature baby when they are pregnant. For these reasons, it is important to have a better understanding of the normal bacteria of the vagina.Some bacteria found in the vagina can not be grown in a laboratory. Our preliminary studies indicate a very wide variety of bacteria in the vagina. Also we have shown there are some differences between African American and Caucasian women. The goal of our study is to study the bacteria in the vagina of normal women using the latest technology. This technology involves study the bacterial DNA present in the normal microbes in the vagina

DETAILED DESCRIPTION:
The normal vaginal bacteria in healthy women of reproductive age plays a key role in preventing successful colonization by "undesirable" organisms including those responsible for bacterial vaginosis, yeast infections, sexually transmitted diseases and urinary tract infections. Our long-term goal is to develop an accurate understanding of the vagina microbial ecosystem in normal, healthy women as an essential prerequisite for comprehending how the normal microflora reduces the risk of acquiring these common vaginal infections.

Four hundred women will be recruited such that there will be equal distribution among four self-declared ethnic groups (Caucasian, African-American, Hispanic and Asian). These groupings were selected based on the original Forney study that identified different distributions supergroups of dominant vaginal microflora between African-American and Caucasian women.

The experimental focus of this proposal is to use a combination of culture-independent methods (T-RFLP of 16S rRNA, 16SrRNA and recA genes sequence analysis and community genomics) to develop tools aimed at advancing our understanding of the composition and role of individual organisms and communities that make up the ecosystems of human vaginas . The specific aims are designed to develop genomic tools for the research and clinical scientific community to study the ecology of the human vaginal microflora

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 12 and 45
* Regular menstrual cycles from 21 to 35 days long
* Normal healthy volunteer
* Negative urine pregnancy test
* Ability to understand and sign informed consent

Exclusion Criteria:

* Used douches, vaginal medications or suppositories, feminine sprays, genital wipes, or contraceptive spermicides in the past 48 hours
* Sexually active in the past 48 hours (involving female genitalia)
* Pregnancy (by history or testing)
* Use of antibiotics or antifungal drugs within the past 30 days
* Have chronic illnesses such as kidney failure, diabetes or HIV/AIDS
* Self-reported vaginal discharge in the past 48 hours
* Currently menstruating
* Currently participating in a drug or treatment clinical research trial
* Received a vaccine within the last 30 days
* Received a vaccine against a bacterial infection
* Currently using NuvaRing for contraception
* Any other condition that in the opinion of the investigator would place the subject in unacceptable risk for participation in the study

Ages: 12 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Asian, African American, Hispanic, or Cauasian women between the ages of 12 to 45 years old
Sampling Method: Non-Probability Sample
Enrollment: 396 (Actual)
Dates: Start 2008-05; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
descriptive analysis of vaginal microbiome | completed

SECONDARY OUTCOMES:
correlate vaginal microbiome to other demographic information, Nugent score and vaginal pH | completed

CONTACTS AND LOCATIONS:
Overall Officials: Jacques Ravel, phD, Principal Investigator — University of Maryland
Locations (3):
- United States (3):
  - Emory University, Atlanta, Georgia
  - Adolescent and Young Adult Center (AYAC),UMB, Baltimore, Maryland
  - Center for Vaccine Development, University of Maryland, Baltimore, Maryland